CLINICAL TRIAL: NCT03517865
Title: International Primary Ciliary Dyskinesia Cohort
Acronym: iPCD
Status: Active, not recruiting | Type: Observational
Sponsor: University of Bern (Other)
Collaborators: European Commission (Other); Swiss National Science Foundation (Other); University of Southampton (Other); Pierre and Marie Curie University (Other); Bar-Ilan University, Israel (Other); University of Padova (Other); University Hospital, Gasthuisberg (Other); Oslo University Hospital (Other); Amsterdam UMC, location VUmc (Other); Royal Brompton & Harefield NHS Foundation Trust (Other); Marmara University (Other); Ruhr University of Bochum (Other); Genetic Disorders of Mucociliary Clearance Consortium (Unknown); Institute of Tuberculosis and Lung Disorders, Rabka Poland (Unknown); University of Sydney (Other); Copenhagen University Hospital, Denmark (Other); University Hospital Muenster (Other); Hannover Medical School (Other); Hospital de Niños R. Gutierrez de Buenos Aires (Other); University of Cyprus (Other); Medical Centre Dr Dragisa Misovic (Unknown); Hacettepe University (Other); University Hospital, Motol (Other); Clinica de neumologia pediatrica Compensar (Unknown); Attikon Hospital (Other); University of Leicester (Other)
Responsible Party: Sponsor
Other Study IDs: iPCD cohort
Record Dates: First submitted 2018-04-05; First posted 2018-05-08 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Primary Ciliary Dyskinesia; Kartagener Syndrome
MeSH Terms: conditions — Ciliary Motility Disorders; Kartagener Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The iPCD Cohort is an international cohort that assembles available retrospective datasets and prospectively newly collected clinical and diagnostic data from patients suffering from primary ciliary dyskinesia (PCD) worldwide, to answer pertinent questions on clinical phenotype, disease severity, prognosis and effect of treatments in patients with this rare multiorgan disease.

DETAILED DESCRIPTION:
The iPCD Cohort was set up under the framework of the European Union (EU) funded 7th Framework Programme (FP7) project Better Experimental Screening and Treatment for Primary Ciliary Dyskinesia (BESTCILIA). The iPCD Cohort is hosted at the Institute of Social and Preventive Medicine at the University of Bern, Switzerland. Research is performed in close collaboration with all data contributors.

Aims:

This combined international dataset allows investigation of PCD epidemiology in a large international study population in order to: 1) describe the spectrum of clinical phenotypes and disease severity in PCD patients by age, sex and time period of diagnosis; 2) describe short-term and long-term prognosis of PCD, looking at important outcomes such as growth, lung function and respiratory failure, bacterial colonisation, hearing loss, fertility, and mortality; and 3) identify predictors of long-term outcomes such as age at diagnosis, clinical phenotype, ultrastructural defects, genotype and clinical care.

Study design:

The iPCD Cohort is an international cohort, combining available data on PCD from national or local registries and clinical or diagnostic databases. All participating centres delivered retrospectively collected data; new centres joining the iPCD Cohort in the future can also participate with retrospectively and prospectively collected data.

What information is collected:

The iPCD Cohort includes retrospectively collected patient data on the following 11 thematic categories: 1) general information, 2) results of diagnostic tests, 3) baseline characteristics, 4) growth and lung function, 5) clinical manifestations, 6) therapy, 7) microbiology, 8) imaging, 9) surgical interventions, 10) neonatal period, and 11) family history.

Study database:

The iPCD Cohort database is web-based, using the Research Electronic Data Capture (REDCap) platform developed at Vanderbilt University. REDCap is widely used in academic research and allows data entry and extraction in various formats.

How to participate:

Centres that wish to participate to the project and contribute data can contact the iPCD Cohort to sign a data delivery agreement. They then will receive a password to access the online software REDCap and they will be able to enter their data directly. They can also upload follow-up data or add additional patients at a later time point.

For further details, contact: pcd@ispm.unibe.ch

Funding:

The setting up of the iPCD Cohort (salaries, consumables and equipment) was funded by the EU FP7 project BESTCILIA (http://bestcilia.eu) and several Swiss funding bodies, including the Lung Leagues of Bern, St Gallen, Vaud, Ticino and Valais and the Milena Carvajal Pro-Kartagener Foundation. Data collection and management at each site was funded according to local arrangements. Most participating researchers and data contributors participate in the European Cooperation in Science and Technology (COST) Action "Better Evidence to Advance Therapeutic options for PCD" (BEAT-PCD) (BM 1407; www.beatpcd.org). Infrastructure is provided for free by the University of Bern, where the data are pooled and stored. The study is currently funded by the Swiss National Science Foundation (320030_173044 and 320030B_192804).

ELIGIBILITY:
Inclusion Criteria:

Patients diagnosed with primary ciliary dyskinesia

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients of all ages diagnosed with PCD, followed in a PCD centre or other specialised clinic or registered in a national registry
Sampling Method: Non-Probability Sample
Enrollment: 3400 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2050-12 (Estimated); Study Completion 2080-12 (Estimated)

PRIMARY OUTCOMES:
Height | every 3 months up to 10 years
  Height z-scores calculated based on available national and international references
BMI | every 3 months up to 10 years
  Body Mass Index (BMI) z-scores calculated based on available national and international references
Lung function measurements | every 3 months up to 10 years
  Spirometric indices, particularly Forced expiratory volume in 1 sec (FEV1) and Forced vital capacity (FVC) z-scores calculated based on Global Lung Function Initiative (GLI) reference values
Diagnostic test results | at diagnosis/ study entry
  Results of performed PCD diagnostic tests including measurement of nasal nitric oxide, electron microscopy findings, beat frequency and pattern.
Clinical symptoms and signs | every 3 months up to 10 years
  Prevalence of reported clinical symptoms at different age groups, including rhinitis, cough, otitis, sinusitis, pneumonia, laterality defects, congenital heart disease and fertility problems.
Microbiology results | every 3 months up to 10 years
  Results of microbiology cultures of respiratory samples (sputum, cough swabs, throat swabs, ear swabs, bronchoalveolar lavage) and information on antibiotic resistance (in positive cultures)
Imaging results | every 3 months up to 10 years
  Radiological findings from sinus and lung imaging tests including x-rays, computed tomography and magnetic resonance imaging

CONTACTS AND LOCATIONS:
Overall Officials: Claudia E Kuehni, Prof, Principal Investigator — University of Bern
Locations (1):
- University of Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Researchers wanting to use the iPCD Cohort dataset can propose a research topic and draft a concept sheet describing the planned analyses and publication. All concept sheets have to be approved by all participating centres contributing data to the proposed analysis under question. After the participating centres agree to contribute their data and sign a publication agreement, the iPCD cohort managing centre (University of Bern) will prepare a partial dataset for the proposed analysis and will work closely with the lead researchers offering methodological input and support. In case additional data is collected to complete the partial dataset for a specific project, this will be added to the iPCD Cohort to enrich it after each project.
  For further details, contact: pcd@ispm.unibe.ch

REFERENCES:
- [Result] Goutaki M, Maurer E, Halbeisen FS, Amirav I, Barbato A, Behan L, Boon M, Casaulta C, Clement A, Crowley S, Haarman E, Hogg C, Karadag B, Koerner-Rettberg C, Leigh MW, Loebinger MR, Mazurek H, Morgan L, Nielsen KG, Omran H, Schwerk N, Scigliano S, Werner C, Yiallouros P, Zivkovic Z, Lucas JS, Kuehni CE; PCD Italian Consortium; Swiss PCD Group; French Reference Centre for Rare Lung Diseases; Genetic Disorders of Mucociliary Clearance Consortium. The international primary ciliary dyskinesia cohort (iPCD Cohort): methods and first results. Eur Respir J. 2017 Jan 4;49(1):1601181. doi: 10.1183/13993003.01181-2016. Print 2017 Jan. PMID 28052956
- [Result] Goutaki M, Halbeisen FS, Spycher BD, Maurer E, Belle F, Amirav I, Behan L, Boon M, Carr S, Casaulta C, Clement A, Crowley S, Dell S, Ferkol T, Haarman EG, Karadag B, Knowles M, Koerner-Rettberg C, Leigh MW, Loebinger MR, Mazurek H, Morgan L, Nielsen KG, Phillipsen M, Sagel SD, Santamaria F, Schwerk N, Yiallouros P, Lucas JS, Kuehni CE; PCD Israeli Consortium; Swiss PCD Group; French Reference Centre for Rare Lung Diseases. Growth and nutritional status, and their association with lung function: a study from the international Primary Ciliary Dyskinesia Cohort. Eur Respir J. 2017 Dec 21;50(6):1701659. doi: 10.1183/13993003.01659-2017. Print 2017 Dec. PMID 29269581
- [Result] Halbeisen FS, Goutaki M, Spycher BD, Amirav I, Behan L, Boon M, Hogg C, Casaulta C, Crowley S, Haarman EG, Karadag B, Koerner-Rettberg C, Loebinger MR, Mazurek H, Morgan L, Nielsen KG, Omran H, Santamaria F, Schwerk N, Thouvenin G, Yiallouros P, Lucas JS, Latzin P, Kuehni CE. Lung function in patients with primary ciliary dyskinesia: an iPCD Cohort study. Eur Respir J. 2018 Aug 23;52(2):1801040. doi: 10.1183/13993003.01040-2018. Print 2018 Aug. PMID 30049738
- [Result] Halbeisen FS, Shoemark A, Barbato A, Boon M, Carr S, Crowley S, Hirst R, Karadag B, Koerner-Rettberg C, Loebinger MR, Lucas JS, Maitre B, Mazurek H, Ozcelik U, Martinu V, Schwerk N, Thouvenin G, Tschanz SA, Yiallouros P, Goutaki M, Kuehni CE. Time trends in diagnostic testing for primary ciliary dyskinesia in Europe. Eur Respir J. 2019 Oct 24;54(4):1900528. doi: 10.1183/13993003.00528-2019. Print 2019 Oct. No abstract available. PMID 31273043
- [Result] Kouis P, Goutaki M, Halbeisen FS, Gioti I, Middleton N, Amirav I; Israeli PCD Consortium; Barbato A; Italian PCD Consortium; Behan L, Boon M, Emiralioglu N, Haarman EG, Karadag B, Koerner-Rettberg C, Lazor R; Swiss PCD Group; Loebinger MR, Maitre B; French Reference Centre for Rare Lung Diseases; Mazurek H, Morgan L, Nielsen KG, Omran H, Ozcelik U, Price M, Pogorzelski A, Snijders D; PCD Italian Consortium; Thouvenin G; French Reference Centre for Rare Lung Diseases; Werner C, Zivkovic Z, Kuehni CE, Yiallouros PK. Prevalence and course of disease after lung resection in primary ciliary dyskinesia: a cohort & nested case-control study. Respir Res. 2019 Sep 18;20(1):212. doi: 10.1186/s12931-019-1183-y. PMID 31533829
- [Result] Goutaki M, Halbeisen FS, Barbato A, Crowley S, Harris A, Hirst RA, Karadag B, Martinu V, Morgan L, O'Callaghan C, Ozcelik U, Scigliano S, Ucros S, Yiallouros P, Schulzke SM, Kuehni CE. Late Diagnosis of Infants with PCD and Neonatal Respiratory Distress. J Clin Med. 2020 Sep 4;9(9):2871. doi: 10.3390/jcm9092871. PMID 32899853
- [Result] Halbeisen FS, Pedersen ESL, Goutaki M, Spycher BD, Amirav I, Boon M, Cohen-Cymberknoh M, Crowley S, Emiralioglu N, Haarman EG, Karadag B, Koerner-Rettberg C, Latzin P, Loebinger MR, Lucas JS, Mazurek H, Morgan L, Marthin J, Pohunek P, Santamaria F, Schwerk N, Thouvenin G, Yiallouros P, Nielsen KG, Kuehni CE. Lung function from school age to adulthood in primary ciliary dyskinesia. Eur Respir J. 2022 Oct 20;60(4):2101918. doi: 10.1183/13993003.01918-2021. Print 2022 Oct. PMID 35301251